CLINICAL TRIAL: NCT07189702
Title: A Randomized Controlled Trial of Behavioral Education and Nutrition Delivery in Women With Metastatic Breast and Endometrial Cancer. (The BEND-MBEC Study)
Brief Title: Plant-Based Nutrition for Breast or Endometrial Cancer
Acronym: BEND-MBEC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Thomas M Campbell, Assistant Professor (Part-Time) - Department of Family Medicine (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00010949
Record Dates: First submitted 2025-09-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Metastatic; Endometrial Cancer Stage IV
Keywords: Metastatic; Metastatic Breast; Metastatic Endometrial; Breast Stage IV; Endometrial Stage IV; Nutrition; Plant-Based Nutrition
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis | interventions — Diet, Plant-Based; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Regular Diet with Cancer-Related Wellness Education and Support
  Interventions: Other: Control
- Whole Food, Plant-Based Diet with Behavioral Education and Support (Experimental): Whole Food, Plant-Based Diet with Behavioral Education and Support
  Interventions: Other: Whole Food, Plant-Based Diet with Behavioral Education and Support

INTERVENTIONS:
Other: Control — Regular Diet with Cancer-Related Wellness Education and Support
  Arms: Control
Other: Whole Food, Plant-Based Diet with Behavioral Education and Support — Whole Food, Plant-Based Diet with Behavioral Education and Support
  Arms: Whole Food, Plant-Based Diet with Behavioral Education and Support

SUMMARY:
This is a randomized controlled trial of a whole food, plant-based (WFPB) dietary intervention among women with metastatic breast or endometrial cancer.

DETAILED DESCRIPTION:
This is a randomized controlled trial of a whole food, plant-based (WFPB) dietary intervention among women with metastatic breast or endometrial cancer. It is designed to explore whether this dietary intervention is sustainable in this population for 26 weeks and whether improvements in quality of life and cardiometabolic health demonstrated in a previous study are sustained. If so, this study will gather information to know whether these benefits translate into reduced overall mortality and cancer markers when compared with a control group that is matched for time and attention but does not implement dietary change. The intervention consists of a whole food plant-based dietary program, group education and individual coaching/visits while the control group gets general wellness group education and individual visits while maintaining their usual diet.

ELIGIBILITY:
Inclusion Criteria: • Female sex (as assigned at birth), aged 18 years or older

* A confirmed diagnosis of endometrial or metastatic breast cancer. All subtypes are eligible
* Treating oncologist approval and expected survival of at least six months
* Undergoing any systemic treatment including hormonal, cytotoxic, targeted monoclonal antibody or small molecule kinase inhibitors or any combination of the above. Women who have active cancer and have been recommended but declined systemic treatment are also eligible.
* Willing to adopt a strict, whole-foods, plant-based diet
* Willing and able to comply with the WFPB protocol for the duration of the study including scheduled testing, Zoom meetings, and office visits
* Able to speak and read English fluently.
* Women with plans for radiation therapy or surgery are also eligible provided that they meet all other eligibility criteria.

Exclusion Criteria: • BMI ≤ 20.0 kg/m2

* Inability to tolerate a normal diet
* Active malabsorption syndrome at time of consent, as determined by study physicians (i.e. Crohn's disease, bowel surgery)
* Any food allergies or intolerances that would interfere with study compliance
* Recent consumption (in the past six months) of a vegan diet
* eGFR < 30 on ≥ two lab tests in the past six months
* Serum potassium > 5.4 in the past six months
* Current insulin or sulfonylurea use
* Current warfarin use (non-vitamin K antagonist allowed)
* High-risk alcohol use (>7 drinks/wk)
* Illicit substance use (not including marijuana)
* Cognitive impairment or psychiatric disorder impairing ability to give consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Dietary Adherence at 13 and 26 Weeks | 13 weeks, 26 weeks
  Dietary adherence is assessed by study personnel using pre-specified criteria. Participants are considered "adherent" if ≥80% of total calories are consumed from 'on-plan' foods. A single adherence score is calculated as the percentage of calories consumed from on-plan foods, averaged over the assessment period. Higher scores indicate greater adherence.
Mean Change in Participant Retention at 13 and 26 Weeks | 13 weeks, 26 weeks
  Retention is calculated as the percentage of consented participants who provide both baseline and post-intervention assessments. Higher percentages indicate better retention in the WFPB dietary intervention.

SECONDARY OUTCOMES:
Mean Change in Disease-Specific Quality of Life - FACT-B at 13 and 26 Weeks | 13 weeks, 26 weeks
  Quality of life is assessed using the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire. Individual item scores are summed to create subscale scores and a total score, with higher scores indicating better quality of life. Mean change from baseline is calculated.
Mean Change in Disease-Specific Quality of Life - FACT-En at 13 and 26 Weeks | 13 weeks, 26 weeks
  Quality of life is assessed using the Functional Assessment of Cancer Therapy - Endocrine (FACT-En) questionnaire. Item responses are summed for subscales and a total score, with higher scores indicating better QOL. Mean change from baseline is evaluated.
Mean Change in Cognitive Dysfunction (FACT-COG) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Cognitive function is measured using the FACT-COG questionnaire. Items are summed to generate a total cognitive dysfunction score. Higher scores indicate greater cognitive function (less dysfunction). Mean change from baseline is calculated to assess improvement or decline.
Mean Change in Cancer-Related Fatigue (BFI) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Fatigue is assessed using the Brief Fatigue Inventory (BFI). Scores for each item range from 0 (no fatigue) to 10 (severe fatigue) and are averaged to obtain a total fatigue score. Lower scores indicate less fatigue. Mean change from baseline is calculated.
Mean Change in General Symptoms (MDASI) at 13 and 26 Week | 13 weeks, 26 weeks
  General symptoms are measured using the MD Anderson Symptom Inventory (MDASI). Items are rated 0-10, with higher scores indicating greater symptom severity. Total symptom burden is calculated by summing items. Mean change from baseline is evaluated to assess improvement.
Overall Survival at Close of Study | End of study (26 weeks)
  Overall survival is defined as the time from study enrollment to death from any cause. Survival status is determined through medical records and follow-up.
Mean Change in Cardiometabolic Marker (Weight) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Weight is collected at each time point, and mean change from baseline is calculated.
Mean Change in Cardiometabolic Marker (Lipids) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Lipids are measured at each time point, and mean change from baseline is calculated.
Mean Change in Cardiometabolic Marker (Blood Pressure) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Blood Pressure is measured at each time point, and mean change from baseline is calculated.
Mean Change in Cardiometabolic Marker (Insulin) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Insulin is measured at each time point, and mean change from baseline is calculated.
Mean Change in Cardiometabolic Marker (Inflammation) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Inflammation is measured at each time point, and mean change from baseline is calculated.
Mean Change in Cardiometabolic Marker (Blood Glucose) at 13 and 26 Weeks Description: | 13 weeks, 26 weeks
  Blood Glucose is measured at each time point, and mean change from baseline is calculated.
Mean Change in Hormonal Marker (IGF1) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Description: IGF1 is measured at each time point, and mean change from baseline is calculated.
Mean Change in Hormonal Marker (sex hormones) at 13 and 26 Weeks | 13 weeks, 26 weeks
  Sex hormones are measured at each time point, and mean change from baseline is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Campbell, MD, Principal Investigator — University of Rochester; Erin K Campbell, MD, MPH, Principal Investigator — University of Rochester

IPD SHARING:
Plan to Share IPD: No